CLINICAL TRIAL: NCT01641224
Title: A Randomized, Double-blind, and Placebo-controlled Study on the Treatments of Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1106E00524
Record Dates: First submitted 2012-05-23; First posted 2012-07-16 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome,; Pinaverium; Herbal medication for IBS,; Tong Xie Yao Fang (Formula for pain and diarrhea)
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — pinaverium; diterpenoid C, Radix curcumae

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TCM (Traditional Chinese medicine) (Active Comparator): Formula for pain and diarrhea, Atractylodes (~10-15g), Paeonia Lactiflora (~15-30g), Tangerine Peel (~10g), Ledebouriella Root (~10g), Radix codonopsitis (~10-15g), Radix curcumae (~10g), Fingered citron (~10g), Tuckahoe (~15g), etc.
  Interventions: Device: Atractylodes; Device: Paeonia Lactiflora; Device: Tangerine Peel; Drug: Ledebouriella Root; Drug: Radix codonopsitis; Drug: Radix curcumae; Drug: Fingered citron; Drug: Tuckahoe
- Pinaverium (Active Comparator)
  Interventions: Drug: Pinaverium
- Placebo (Placebo Comparator): Placebo is blindly given to patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pinaverium — To test the effectiveness and safety of the formula for pain and diarrhea, we will randomly assign patients into one 3 groups: Pinaverium, TCM (Formula for pain and diarrhea) group, and placebo group, and treat them accordingly.
  Arms: Pinaverium
Device: Atractylodes — Atractylodes (~10-15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Device: Paeonia Lactiflora — Paeonia Lactiflora (~15-30g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Device: Tangerine Peel — Tangerine Peel (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Ledebouriella Root — Ledebouriella Root (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Radix codonopsitis — Radix codonopsitis (~10-15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Radix curcumae — Radix curcumae (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Fingered citron — Fingered citron (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Tuckahoe — Tuckahoe (15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Placebo — Placebo is blindly given to patients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the efficacy and safety of pinaverium and an herbal medication for irritable bowel syndrome (IBS). Pinaverium has been in many countries, but there is no randomized, double-blind, large sample size, and placebo-controlled study on this medication yet. Tong Xie Yao Fang (Formula for pain and diarrhea) is a historically and contemporarily used traditional Chinese medicine that can be used for IBS. The hypothesis is that the two remedies are effective and safe for IBS treatment when tested by modern clinical standards and criteria.

DETAILED DESCRIPTION:
Pinaverium bromide (pinaverium), an antispasmodics, is one of the most commonly used IBS medication worldwide. However, original clinical studies on pinaverium are scarce. Only five original clinical studies from Europe, one from Latin America, and one from Asian were found. These studies were single-centered and small sample sized (19 - 53 IBS patients) studies.

Tong Xie Yao Fang has long been used in China. Its efficacy and safety has not been evaluated by modern scientific method.

This study is designed to evaluate the efficacy and safety of pinaverium and Tong Xie Yao Fang for IBS treatment in a double-blind, randomized, and large sample size clinical trial using placebo as a control.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old age group, male and female
* In accordance with the above Western medicine Rome III standards.
* In accordance with the above description of Deficient Spleen Qi and Liver Qi Stagnation
* Informed consent for treatment
* No change in appetite during treatments periods

Exclusion Criteria:

* Pregnant or lactation female patients, and Fertility male patients
* Present digestive system disease within current three months
* Take IBS medicines within ten days prior to treatment or during treatment
* Take depression medicine within ten days prior to treatment or during treatment
* Take pain reliever medicine within ten days prior to treatment or during treatment
* Have serious primary heart, liver, kidney, lung and blood system diseases, asthma, and Lung and liver dysfunction patients
* If an emergency occurs; a physician terminates the treatment
* Cannot comply with the rules and cannot cooperate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The relief of irritable bowel syndrome symptoms was used to measure the effectiveness of the drugs | TCM group: 4 weeks. Pinaverium: 4 weeks. Placebo: 4 weeks.
  The parameters used to evaluate the effectiveness of the drugs included i) Abdominal pain (0 = no pain, 1 = mild pain, 2 = moderate pain, 3 = severe pain); ii) Frequency of the pain (# of pains per day); iii) Abdominal discomfort (0 = No discomfort,1 = mild,2 = moderate,3 = severe); iv) Frequency of discomfort (# of discomfort per day); v) # of stools per day; vi) Form (appearance) of stool (0 = Normal,1 = soft pieces with clear-cut edges,2 = mushy,3 = watery)

SECONDARY OUTCOMES:
The side effect associated with the treatments | TCM group: 4 weeks. Pinaverium: 4 weeks. Placebo: 4 weeks.
  The following will be documented: constipation, headache, dizzy, hypertension, chest pain, abdominal pain, flatus, anxiety, insomnia, nausea, fever, fatigue, muscle pain, urinary infection, respiratory tract infection, Others.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Xiao, Ph.D., Principal Investigator — University of Minnesota
Locations (4):
- China (4):
  - Second Jiangsu Provincial Hospital of Traditional Chinese Medicine affiliated to Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine affiliated to Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Beijing Xuanwu Hospital of Traditional Chinese Medicine affiliated to Capital Medical University., Beijing
  - Shanghai First People's Hospital affiliated to Shanghai Tiao Tong University, Shanghai

REFERENCES:
- [Derived] Wang Y, Fan H, Qi X, Lai Y, Yan Z, Li B, Tang M, Huang D, Li Z, Chen H, Zhu Q, Luo C, Chen X, Fen J, Jiang Z, Zheng L, Liu X, Tang Q, Zuo D, Ye J, Yang Y, Huang H, Tang Z, Lu W, Xiao J; Pharm D for the China Irritable Bowel Syndrome Consortium. Are personalized tongxie formula based on diagnostic analyses more effective in reducing IBS symptoms?-A randomized controlled trial. Complement Ther Med. 2018 Oct;40:95-105. doi: 10.1016/j.ctim.2018.07.002. Epub 2018 Aug 8. PMID 30219477
- [Derived] Fan H, Zheng L, Lai Y, Lu W, Yan Z, Xiao Q, Li B, Tang M, Huang D, Wang Y, Li Z, Mei Y, Jiang Z, Liu X, Tang Q, Zuo D, Ye J, Yang Y, Huang H, Tang Z, Xiao J; China Irritable Bowel Syndrome Consortium. Tongxie Formula Reduces Symptoms of Irritable Bowel Syndrome. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1724-1732. doi: 10.1016/j.cgh.2017.06.026. Epub 2017 Jun 17. PMID 28634136
- [Derived] Zheng L, Lai Y, Lu W, Li B, Fan H, Yan Z, Gong C, Wan X, Wu J, Huang D, Wang Y, Mei Y, Li Z, Jiang Z, Liu X, Ye J, Yang Y, Huang H, Xiao J. Pinaverium Reduces Symptoms of Irritable Bowel Syndrome in a Multicenter, Randomized, Controlled Trial. Clin Gastroenterol Hepatol. 2015 Jul;13(7):1285-1292.e1. doi: 10.1016/j.cgh.2015.01.015. Epub 2015 Jan 26. PMID 25632806